CLINICAL TRIAL: NCT05068245
Title: Music to Reduce Patient Reported Pain During Intrauterine Device (IUD) Placement in the Office
Acronym: MIUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Glenmarie Matthews, MD, Assistant Professor, Family Planning Specialist, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020000698
Record Dates: First submitted 2021-09-02; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Pain, Acute; Anxiety
Keywords: Intrauterine Devices
MeSH Terms: conditions — Acute Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The intervention being tested is music. Patients will receive either routine pain control measures only (control group) or routine pain control measures and music (treatment group). Routine pain control will include instructions to take ibuprofen 600 mg 30 minutes prior to the procedure. These instructions will be given to all participants. It will be noted whether patients actually take ibuprofen or not by the study staff. Patients randomized to receive music in addition to routine pain control measures, will listen to preselected classical music.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine pain control (No Intervention): The routine pain control group will receive instructions to take ibuprofen 600 mg 30 minutes prior to the procedure. These instructions will be given to all participants.
- Routine pain control plus music (Experimental): Patients randomized to receive music in addition to routine pain control measures, will be instructed to take ibuprofen 600 mg 30 minutes prior to the procedure. These instructions will be given to all participants. Preselected classical music will be played for this group throughout the procedure.
  Interventions: Behavioral: Preselected classical music

INTERVENTIONS:
Behavioral: Preselected classical music — Preselected classical music
  Other Names: Music
  Arms: Routine pain control plus music

SUMMARY:
This study seeks to determine if music reduces pain and anxiety in comparison to routine pain control measures alone during insertion of intrauterine contraceptive devices (Mirena, Paragard)

DETAILED DESCRIPTION:
This will be a randomized control trial conducted in the gynecology clinic inside Robert Wood Johnson University Hospital (RWJ) and the offices of Rutgers Medical Group Obstetrics and Gynecology (RMG). A family planning attending alone at RMG or accompanied by obstetrics and gynecology (Ob/Gyn) residents at RWJ will perform all IUD insertions during this study period. Patients scheduled for an IUD, either the Mirena® (levonorgestrel-releasing intrauterine system 52 mg) or Paragard® (intrauterine copper contraceptive), at both locations will be instructed to take ibuprofen 30 minutes prior to their procedure.

Enrollment will occur during all weekdays at both RWJ and RMG. Eligible women will be enrolled if they are willing to be randomized. Written consent will be obtained from each participant.

After the consent process is completed, the patients will complete a survey which includes their demographic information, if they are currently menstruating, and their pregnancy history while sitting in the waiting room. The patient will also complete a 10 point visual analog scale (VAS) to report her baseline pain and a State Trait Anxiety Inventory (STAI). Vital signs will be recorded with an automated machine.

Participants will then be randomized to routine pain control measures or routine pain control measures plus music. Randomization will be completed by the study staff, who will open sequentially numbered, sealed, opaque envelopes. Allocation will be in a 1:1 ratio. Routine pain control will include instructions to take ibuprofen 600 mg 30 minutes prior to the procedure. These instructions will be given to all participants. It will be noted whether patients actually take ibuprofen or not by the study staff. Patients randomized to receive music in addition to routine pain control measures, will be given a headset that will be plugged into the PI phone to play the preselected classical music. Patients will control the volume. Control group participants also will receive a headset. The headsets will not be noise cancelling.

A study staff member will be present in the room throughout the duration of the procedure in addition to the physician performing the actual insertion of the IUD. This study staff member will complete a procedure information sheet including vitals, type of IUD inserted, and the VAS and STAI at several points of the procedure (immediately prior to the procedure, point of speculum insertion, point of tenaculum placement, point of IUD insertion, and 5 minutes post-procedure).

ELIGIBILITY:
Inclusion Criteria:

* Women who have an appointment for IUD insertion at either RWJ or RMG
* Women who are able to read and write in English or Spanish
* Age equal to or greater than 18 years

Exclusion Criteria:

* Contraindications to IUD placement: Active pelvic infection, pregnancy, known distortion of uterine cavity, Wilson's disease (Paragard® only), breast cancer (Mirena® only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Pain to be reported via a 10 point visual analog scale (VAS) | Immediately prior to the procedure, at the point of speculum insertion, at the point of tenaculum placement, at the point of intrauterine device insertion, and five minutes post-procedure
  Pain will be reported via a 10 point visual analog scale (VAS), from a score of 0 to 10 with 0 being no pain (better outcome) and 10 being the most pain (worse outcome).
Pain to be reported via a 10 point visual analog scale (VAS) | At the point of speculum insertion, at the point of tenaculum placement, at the point of intrauterine device insertion, and five minutes post-procedure
  Pain will be reported via a 10 point visual analog scale (VAS), from a score of 0 to 10 with 0 being no pain (better outcome) and 10 being the most pain (worse outcome).
Pain to be reported via a 10 point visual analog scale (VAS) | At the point of tenaculum placement, at the point of intrauterine device insertion, and five minutes post-procedure
  Pain will be reported via a 10 point visual analog scale (VAS), from a score of 0 to 10 with 0 being no pain (better outcome) and 10 being the most pain (worse outcome).
Pain to be reported via a 10 point visual analog scale (VAS) | At the point of intrauterine device insertion, and five minutes post-procedure
  Pain will be reported via a 10 point visual analog scale (VAS), from a score of 0 to 10 with 0 being no pain (better outcome) and 10 being the most pain (worse outcome).
Pain to be reported via a 10 point visual analog scale (VAS) | Five minutes post-procedure
  Pain will be reported via a 10 point visual analog scale (VAS), from a score of 0 to 10 with 0 being no pain (better outcome) and 10 being the most pain (worse outcome).

SECONDARY OUTCOMES:
Anxiety to be reported via the State Trait Anxiety Inventory (STAI) | Anxiety will be recorded immediately prior to the procedure and five minutes post-procedure
  Anxiety will be reported via the State Trait Anxiety Inventory (STAI), which is scale with a minimum value of 10 (better outcome) and a maximum value of 40 (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: AMY J PATEL, MD, Study Director — Rutgers, The State University of New Jersey; Glenmarie Matthews, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: The data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. To gain access, data requestors should direct proposals to ajp323@rwjms.rutgers.edu.

REFERENCES:
- [Background] Abdelhakim AM, Samy A, Abbas AM. Effect of music in reducing patient anxiety during colposcopy: A systematic review and meta-analysis of randomized controlled trials. J Gynecol Obstet Hum Reprod. 2019 Dec;48(10):855-861. doi: 10.1016/j.jogoh.2019.07.007. Epub 2019 Jul 2. PMID 31276848
- [Background] Practice Bulletin No. 186 Summary: Long-Acting Reversible Contraception: Implants and Intrauterine Devices. Obstet Gynecol. 2017 Nov;130(5):1173-1175. doi: 10.1097/AOG.0000000000002394. PMID 29064966
- [Background] Akers AY, Steinway C, Sonalkar S, Perriera LK, Schreiber C, Harding J, Garcia-Espana JF. Reducing Pain During Intrauterine Device Insertion: A Randomized Controlled Trial in Adolescents and Young Women. Obstet Gynecol. 2017 Oct;130(4):795-802. doi: 10.1097/AOG.0000000000002242. PMID 28885425
- [Background] Callahan DG, Garabedian LF, Harney KF, DiVasta AD. Will it Hurt? The Intrauterine Device Insertion Experience and Long-Term Acceptability Among Adolescents and Young Women. J Pediatr Adolesc Gynecol. 2019 Dec;32(6):615-621. doi: 10.1016/j.jpag.2019.08.004. Epub 2019 Aug 8. PMID 31401254
- [Background] Chor J, Bregand-White J, Golobof A, Harwood B, Cowett A. Ibuprofen prophylaxis for levonorgestrel-releasing intrauterine system insertion: a randomized controlled trial. Contraception. 2012 Jun;85(6):558-62. doi: 10.1016/j.contraception.2011.10.015. Epub 2011 Dec 15. PMID 22176793
- [Background] Guerrero JM, Castano PM, Schmidt EO, Rosario L, Westhoff CL. Music as an auxiliary analgesic during first trimester surgical abortion: a randomized controlled trial. Contraception. 2012 Aug;86(2):157-62. doi: 10.1016/j.contraception.2011.11.017. Epub 2012 Jan 10. PMID 22240180
- [Background] Lee JH. The Effects of Music on Pain: A Meta-Analysis. J Music Ther. 2016 Winter;53(4):430-477. doi: 10.1093/jmt/thw012. Epub 2016 Oct 19. PMID 27760797

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT05068245/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT05068245/ICF_001.pdf